CLINICAL TRIAL: NCT05442775
Title: A Phase 3, Open-Label Extension of COURAGE-ALS (CY 5031)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The DMC recommended the trial be discontinued due to futility following a planned second interim analysis of the parent trial (CY 5031).
Sponsor: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CY 5032; 2021-004727-33 (EudraCT Number)
Record Dates: First submitted 2022-06-16; First posted 2022-07-05 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-07

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; ALS; CK-2127107; Reldesemtiv
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — reldesemtiv

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Reldesemtiv 300 mg twice daily (Experimental): Patients in this arm take 1 reldesemtiv 300 mg oral tablet twice a day for a 600 mg total daily dose (TDD). Participants who had been down titrated during the parent trail take 150 mg by mouth twice a day.
  Interventions: Drug: Reldesemtiv

INTERVENTIONS:
Drug: Reldesemtiv — Oral tablet

SUMMARY:
The purpose of this study is to assess the long-term safety and tolerability of reldesemtiv in patients with ALS who have successfully completed dosing in the Phase 3 clinical trial, CY 5031 (also known as COURAGE-ALS)

DETAILED DESCRIPTION:
CY 5032 is an open-label extension (OLE) study of the selective fast skeletal muscle troponin activator, reldesemtiv, in patients with ALS who finished dosing (through Week 48) in CY 5031 (COURAGE-ALS). Approximately 400 patients from the sites that participated in CY 5031 are expected to be enrolled in the open-label extension, CY 5032.

Following enrollment, patients will continue dosing with reldesemtiv, 300 mg twice a day for a 600 mg total daily dose (TDD) for a period of 48 weeks.

At the end of 48 weeks, patients may transition to a reldesemtiv Managed Access Program (MAP) if the treating physician agrees to participate in the program.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and willing to sign an ICF and willing to comply with all study procedures and restrictions for the duration specified in the Schedule of Activities. If non-written consent is given, a Legal Designee of the patient must sign the ICF form.
* Completed dosing in CY 5031

Exclusion Criteria:

* Has taken investigational study drug (other than reldesemtiv) prior to dosing, within 30 days or five half-lives of the prior agent, whichever is greater
* Presence on Day 1 of any medically significant cardiac, pulmonary, gastrointestinal, musculoskeletal, or psychiatric illness that might interfere with the patient's ability to comply with study procedures or that might confound the interpretation of clinical safety or efficacy data.
* Use of a strong cytochrome P450 (CYP) 3A4 inhibitor within 7 days prior to first dose of reldesemtiv in CY 5032 or a strong CYP3A4 inducer within 14 days prior to first dose of reldesemtiv in CY 5032
* Use of a medication that is an OCT1/OCT2 substrate within 7 days prior to first dose of reldesemtiv in CY 5032
* Currently participating in another trial, managed access program, open label extension, early access program, or through the right to try act is receiving an investigational drug or received an investigational drug or device within 30 days (or 5 half-lives for drugs, whichever is longer) prior to Day 1. Patients also cannot be taking outside of a clinical trial certain investigational drugs (which includes drugs, supplements, and nutraceuticals) that are currently being studied or have been studied for the treatment of ALS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2022-08-04 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cytokinetics MD, Study Chair — Scientific Leadership at Cytokinetics
Locations (41):
- United States (21):
  - St. Joseph's Hospital & Medical Center - Barrow Neurological Institute, Phoenix, Arizona
  - University of California Irvine - ALS & Neuromuscular Center, Orange, California
  - California Pacific Medical Center - Forbes Norris MDA/ALS Research Center, San Francisco, California
  - University of Colorado Hospital Anschutz Outpatient Pavilion, Aurora, Colorado
  - George Washington Medical Faculty Associates, Washington D.C., District of Columbia
  - University of Florida, Jacksonville, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of South Florida - Carol and Frank Morsani Center for Advanced Health Care, Tampa, Florida
  - Indiana University IU Health Neuroscience Center, Indianapolis, Indiana
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins Outpatient Center, Baltimore, Maryland
  - Michigan Medicine, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Neurology Associates, Lincoln, Nebraska
  - Hospital for Special Surgery, New York, New York
  - SUNY Upstate Medical University Institute for Human Performance, Syracuse, New York
  - Atrium Health Neuroscience Institute, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Texas Neurology, P.A., Dallas, Texas
  - Virginia Commonwealth University, Henrico, Virginia
  - Froedtert Hospital - Department of Neurology, Milwaukee, Wisconsin
- Australia (3):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Royal Brisbane and Women's Hospital, Neurology Department, Herston, Queensland
  - The Perron Institute, Nedlands
- Uz Leuven Gasthuisberg Department of Neurology, Leuven, Belgium
- Canada (9):
  - University of Calgary - Heritage Medical Research Clinic, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Stan Cassidy Centre for Rehabilitation, Fredericton, New Brunswick
  - McMaster University, Hamilton, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
  - University of Saskatchewan, Saskatoon, Saskatchewan
  - CHU de Quebec-Universite Laval, Québec
- RSCI Education and Research Center Beaumount Hospital, Dublin, Ireland
- Italy (2):
  - IRCCS Istituto Auxologico Italiano Ospedale San Luca U.O. Neurologia e Stroke Unit, Milan
  - AOU Citta della Salute e della Scienza di Torino Universita degli Studi di Torino P.O. Mollinette - Dipartimento de Neuroscienze "Rita Levi Montalcini", Torino
- UMC Utrecht Department of Neurology, ALS Center, Utrecht, Netherlands
- Spain (2):
  - Hospital San Rafael, Madrid
  - Hospital Universitario y Politecnico La Fe, Valencia
- Studieenheten, Akademiskt Specialistcentrum, Stockholm, Sweden

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 41 trial centers in North America, Europe, and Australia. The first participant was enrolled on 04 Aug 2022 and the last participant completed on 07 Jun 2023.
Pre-assignment Details: A total of 71 participants who were previously enrolled in the double-blind placebo-controlled CY 5031 parent trial were enrolled in this trial and received at least one dose of reldesemtiv.
Groups:
- Reldesemtiv: Participants in this arm take 1 reldesemtiv 300 mg oral tablet twice a day for a 600 mg total daily dose (TDD)
  Reldesemtiv: Oral tablet
Period: Overall Study
Arm/Group | Reldesemtiv
Started | 71
Completed | 0 (Trial was prematurely terminated by the Sponsor.)
Not Completed | 71
Not completed — Trial terminated | 61
Not completed — Lack of Efficacy | 4
Not completed — Withdrawal by Subject | 4
Not completed — Death | 1
Not completed — Participant removed at Sponsor request | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Arm/Group | Reldesemtiv
Number analyzed (Participants) | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (11.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 69
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 65
  Other | 3
  Asian | 2
  Black or African American | 1
Region of Enrollment [Count of Participants; unit: Participants]
  North America | 53
  Europe | 10
  Australia | 8
Time Since ALS Diagnosis at Screening in CY 5031 [Mean (Standard Deviation); unit: months] | 17.9 (4.69)
Percent Predicted Forced Vital Capacity [Mean (Standard Deviation); unit: percent predicted] | 70.6 (22.76)
ALSFRS-R Total Score [Mean (Standard Deviation); unit: scores on a scale] — ALSFRS-R = Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised. ALSFRS-R total score range is from 0 to 48. A score of 48 reflects normal function.
  scores on a scale | 29.8 (8.47)

OUTCOME MEASURES:

1. Primary Outcome: Long-term Safety and Tolerability
Description: Incidence of treatment-emergent adverse events
Time Frame: Baseline to Week 34 (time the study was terminated prematurely)
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Reldesemtiv
Number analyzed (Participants) | 71
Participants | 39

2. Secondary Outcome: Long-term Effect of Reldesemtiv on ALSFRS-R Functional Outcomes
Description: Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) total scores. ALSFRS-R total score range is from 0 to 48. A score of 48 reflects normal function.
Time Frame: Baseline to Week 32 (last timepoint before study was terminated prematurely)
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reldesemtiv
Number analyzed (Participants) | 71
score on a scale
  Week 12: number analyzed (Participants) | 47
  Week 12 | 29.5 (9.04)
  Week 24: number analyzed (Participants) | 20
  Week 24 | 27.4 (11.86)
  Week 32: number analyzed (Participants) | 9
  Week 32 | 26.6 (13.96)

ADVERSE EVENTS:
Time Frame: up to 34 weeks (time the study was terminated prematurely)
Arm/Group | Reldesemtiv
All-Cause Mortality (participants affected / at risk) | 5/71
Serious Adverse Events (participants affected / at risk) | 11/71
Other Adverse Events (participants affected / at risk) | 27/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reldesemtiv (N=71)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Assisted suicide (Psychiatric disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 1 (1)
Klebsiella urinary tract infection (Infections and infestations) | 1 (1)
Metapneumovirus infection (Infections and infestations) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reldesemtiv (N=71)
Diarrhoea (Gastrointestinal disorders) | 7 (7)
Constipation (Gastrointestinal disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 4 (4)
Urinary tract infection (Infections and infestations) | 5 (5)
Fall (Injury, poisoning and procedural complications) | 5 (5)

LIMITATIONS AND CAVEATS:
Based on interim analysis results of the Phase 3 parent trial CY 5031 which met the criteria for futility in participants with ALS, CY 5032 was prematurely terminated on 31 March 2023.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-12-16): https://cdn.clinicaltrials.gov/large-docs/75/NCT05442775/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-16): https://cdn.clinicaltrials.gov/large-docs/75/NCT05442775/SAP_001.pdf